CLINICAL TRIAL: NCT00786643
Title: Phase II Study of Gamma Interferon (IFN-γ) Added to Bolus + Infusional 5-Fluorouracil (5-FU) and Leucovorin (LV) +/- Bevacizumab (BV) in Metastatic Colorectal Carcinoma
Brief Title: Study of Gamma Interfereon in Metastatic Colorectal Carcinoma
Acronym: GFL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Accelerated Community Oncology Research Network (Other)
Collaborators: InterMune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WITMMCC0301
Record Dates: First submitted 2008-11-03; First posted 2008-11-06 (Estimated); Results first posted 2012-02-22 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Colorectal Cancer
Keywords: Gamma Interferon; 5-FU; LV
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Fluorouracil; Leucovorin; Interferon-gamma; interferon gamma-1b; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stratum 1 (Experimental): Patients in stratum 1 have not received prior chemotherapy in the metastatic setting.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin (LV); Drug: Gamma-Interferon-1b (IFN-γ); Drug: Bevacizumab
- Stratum 2 (Experimental): Patients in stratum 2 have received 1-2 prior chemotherapy regimens in the metastatic setting.
  Interventions: Drug: 5-Fluorouracil; Drug: Leucovorin (LV); Drug: Gamma-Interferon-1b (IFN-γ)

INTERVENTIONS:
Drug: 5-Fluorouracil — 5-FU bolus was administered at 400mg/m^2 on day 1 and day 2 of each cycle. 5-FU at 600 mg/m^2 infusion was administered over 22 hours on day 1 and day 2 of each cycle.
  Other Names: Fluororacil; 5-FU
Drug: Leucovorin (LV) — Leucovorin 200mg/m^2 was administered over 2 hours on day 1 and day 2 of each cycle.
  Other Names: leucovorin calcium; folinic acid
Drug: Gamma-Interferon-1b (IFN-γ) — Gamma-Interferon 150 mcg/m^2 was administered by subcutaneous injection on day 1 of each cycle immediately before treatment with 5-FU and LV, and on day 3 of each cycle immediately after treatment with 5-FU and LV.
  Other Names: Gamma-Interferon-1b; Gamma-Interferon; Actimmune
Drug: Bevacizumab — Bevacizumab 5mg/kg was only added to the treatment regimen of patients in stratum 1 who demonstrated stable disease on imaging repeated prior to the 5th cycle of treatment. Bavacizumab was administered on day 4 of each cycle.
  Other Names: Avastin
  Arms: Stratum 1

SUMMARY:
The purpose of this study is to evalute the response and toxicity of metastatic colorectal cancer patients to the regimen of gamma interferon added to bolus and infusional 5-fluorouracil and leucovorin (GFL) with or without bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic colorectal cancer, histologically or cytologically confirmed
* Age 18 or greater
* Adequate hematologic function (ANC > 1500, hemoglobin > 10 g/dl, platelet count > 100,000)
* Adequate hepatic parameters (bilirubin < 2.0, Alk. Phos < 5 times normal, ALT < 5 times normal)
* Adequate renal function (creatinine < 2.0)
* Performance status ECOG 0-2
* 0-2 prior lines of chemotherapy for metastatic colorectal cancer are allowed. Prior 5-FU/LV or capecitabine allowed either in the adjuvant setting, or in the metastatic setting or both.
* Absence of other serious concurrent medical illnesses
* Evaluable or measurable disease for phase I; measurable disease only for phase II

Exclusion Criteria:

* Histologies other than adenocarcinoma
* Previous grade 4 toxicity to 5-FU +/- LV or capecitabine
* Uncontrolled brain metastases
* Chronic diarrhea (greater than five bowel movements per day)
* Previous chemotherapy or radiation therapy less than 4 weeks prior to study day 1 (less than 6 weeks for chemotherapy with Mitomycin or nitrosoureas)
* Major surgery within 2 weeks before study entry
* Known allergic sensitivity to leucovorin
* Prior exposure to IFN-γ
* Previous hematopoietic growth factor (e.g. epoetin alfa or darbepoietin less than 2 weeks prior to study day 1)
* Pregnancy or breast feeding. Women of child-bearing potential must have a negative pregnancy test before the first dose.
* Other co-existing malignancies or malignancies diagnosed within the last 5 years, with the exception of basal cell carcinoma or cervical cancer in situ
* Inability to provide written and informed consent
* Uncontrolled hypertension
* History of deep venous thrombosis or CVA
* Prior exposure to bevacizumab
* Proteinuria > 500 mg/24 hr

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2006-02; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lee Schwartzberg, MD, Study Chair — Vector Oncology
Locations (1):
- The West Clinic, Memphis, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One community oncology research site in the US within the ACORN Network participated in this study. Phase II enrollment started in February 2006 and was closed in December 2008.
Pre-assignment Details: Informed consent was obtained from all subjects. All subjects underwent a screening period during which pre-study assessments were completed. Subjects were assigned to a stratum, based on whether or not they had received previous treatment in the metastatic setting, at the time of study enrollment.
Period: Overall Study
Arm/Group | Stratum 1 | Stratum 2
Started | 20 | 28
Completed | 20 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stratum 1 | Stratum 2 | Total
Number analyzed (Participants) | 20 | 28 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 19 | 30
  >=65 years | 9 | 9 | 18
Age Continuous [Mean (Standard Deviation); unit: years] | 62.75 (12.05) | 62.32 (10.13) | 62.50 (10.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 15 | 24
  Male | 11 | 13 | 24
Region of Enrollment [Number; unit: participants]
  United States | 20 | 28 | 48

OUTCOME MEASURES:

1. Primary Outcome: Best Response (BR)
Description: BR is recorded from start of treatment until progressive disease (PD). Imaging was repeated by same technique after every 4 cycles of treatment. Response was evaluated per Response Evaluation Criteria In Solid Tumors (RECIST) guidelines version 1.0. Per RECIST v1.0 and CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of longest diameter of target lesions; Stable Disease (SD), neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; PD, increase in existing lesions or new lesions.
Time Frame: After every 4 cycles of treatment (approximately every 56 days for up to about 280 days)
Population: The best response is the best response recorded from the start of treatment until disease progression. Imaging was repeated by same technique after every 4 cycles of treatment. Subjects in both strata were evaluated for this outcome.
Measure: Number; unit: Participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 20 | 28
Participants
  Complete response (CR) | 0 | 0
  Partial response (PR) | 6 | 3
  Stable disease (SD) | 7 | 15
  Progressive disease (PD) | 6 | 6
  Not evaluable (NE) | 1 | 4

2. Secondary Outcome: Early Response Rate (RR) (Stratum 1 Only)
Description: Early RR evaluated in stratum 1 to see if bevacizumab (bev) would be added to GFL treatment (tx). Patients with stable disease (SD) pre 5th cycle of tx had bev added. Response was evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) version 1.0. Per RECIST and CT scan: Complete Response (CR), disappearance of all target lesions; Partial Response (PR), >=30% decrease in sum of longest diameter (LD) of target lesions; SD, neither sufficient shrinkage in sum of LD of target lesions to be PR nor increase of >=20%; Progressive Disease (PD), increase in existing lesions or new lesions.
Time Frame: After 4 cycles of treatment (approximately 56 days)
Population: Prior to the 5th cycle of treatment, early response rate was evaluated in patients in stratum 1 to assess whether bevacizumab would be added to the GFL treatment regimen. Stratum 1 patients with SD at this time point will have bevacizumab added to the regimen. Subjects in stratum 2 were not evaluated for this outcome.
Measure: Number; unit: Participants
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 20 | 0
Participants
  Complete response (CR) | 0 |
  Partial response (PR) | 5 |
  Stable disease (SD) | 7 |
  Progressive disease (PD) | 6 |
  Not evaluable (NE) | 2 |

3. Secondary Outcome: Time to Progression
Description: Patients were censored if they did not progress, stopped particiaption due to an adverse event, or withdrew consent following the start of study treatment. Response was evaluated by Response Evaluation Criteria In Solid Tumors (RECIST) guidelines version 1.0. Per RECIST v1.0, Progressive Disease (PD) is defined as a measurable increase in smallest diameter of any target or non-target lesion, or the appearance of new lesions, since baseline.
Time Frame: From date of study treatment start until date of first documented progression or date of death from any cause, whichever came first, assessed up to 15 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Stratum 1 | Stratum 2
Number analyzed (Participants) | 20 | 28
Months | 5.5263 [3.03 to 6.45] | 3.9145 [3.75 to 7.37]

ADVERSE EVENTS:
Time Frame: Adverse events were collected beginning on day 1 of study treatment until one month after the end of study treatment (approximately every 14 days for up to 310 days).
Description: Systematic Assessment - subjects were assessed for adverse events on day 1 of each cycle (every other week) by either the research coordinator, treating physician, or other appropriate sub-investigator.
Arm/Group | Stratum 1 | Stratum 2
Serious Adverse Events (participants affected / at risk) | 2/20 | 5/27
Other Adverse Events (participants affected / at risk) | 19/20 | 26/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 (N=20) | Stratum 2 (N=27)
Anemia (Blood and lymphatic system disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 2
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Suprapubic pain (General disorders) | 1 | 0
Abdominal infection (Infections and infestations) | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1
Urine output decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stratum 1 (N=20) | Stratum 2 (N=27)
Anaemia (Blood and lymphatic system disorders) | 4 | 3
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 6 | 12
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Congestive cardiomyopathy (Cardiac disorders) | 1 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 0
Lacrimation increased (Eye disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 4 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 9
Dry mouth (Gastrointestinal disorders) | 4 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 3
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 10 | 5
Oral pain (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 2
Vomiting (Gastrointestinal disorders) | 5 | 1
Asthenia (General disorders) | 4 | 2
Chest pain (General disorders) | 0 | 3
Chills (General disorders) | 3 | 2
Face oedema (General disorders) | 0 | 1
Fatigue (General disorders) | 9 | 15
Gait disturbance (General disorders) | 1 | 0
Influenza like illness (General disorders) | 1 | 1
Malaise (General disorders) | 0 | 1
Mucosal inflammation (General disorders) | 2 | 2
Oedema (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 2 | 3
Pain (General disorders) | 4 | 1
Pyrexia (General disorders) | 6 | 3
Hypersensitivity (Immune system disorders) | 1 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1
Sinusitis (Infections and infestations) | 0 | 2
Tooth abscess (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 3
Urinary tract infection (Infections and infestations) | 4 | 3
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Incision site pain (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0
Blood magnesium decreased (Investigations) | 1 | 0
Blood pressure decreased (Investigations) | 1 | 0
Body temperature (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 2 | 0
Platelet count decreased (Investigations) | 0 | 1
Prothrombin time prolonged (Investigations) | 1 | 0
Weight decreased (Investigations) | 2 | 3
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Fluid intake reduced (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2
Burning sensation (Nervous system disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 4 | 3
Memory impairment (Nervous system disorders) | 1 | 0
Mental impairment (Nervous system disorders) | 0 | 1
Neuropathy peripheral (Nervous system disorders) | 2 | 2
Paraesthesia (Nervous system disorders) | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0
Sinus headache (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 0 | 2
Insomnia (Psychiatric disorders) | 3 | 3
Restlessness (Psychiatric disorders) | 0 | 1
Nocturia (Renal and urinary disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 3
Proteinuria (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Scrotal irritation (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 1
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 2 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 3 | 1
Hypertension (Vascular disorders) | 3 | 1
Hypotension (Vascular disorders) | 3 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Enrollment to stratum 1 was closed early due to difficulty accruing the required number of patients in this stratum.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If the Investigator wishes to make a submission for a presentation or publication, the Investigator shall submit all such materials to InterMune at least 60 days prior to the date on which such submission is proposed to be made, and InterMune shall provide timely review of such materials. InterMune may cause the presentation or submission to be delayed for up to 60 additional days if patentable material or proprietary information is identified.